CLINICAL TRIAL: NCT03351166
Title: A Single Arm, Multicenter Study to Investigate the Efficacy and Safety of Oral Molidustat in Dialysis Subjects With Renal Anemia Who Are Not Treated With Erythropoiesis-Stimulating Agents (ESAs)
Brief Title: A Study of Molidustat for Correction of Renal Anemia in Dialysis Subjects
Acronym: MIYABI HD-C
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19351
Record Dates: First submitted 2017-11-20; First posted 2017-11-22 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Anemia; Renal Insufficiency, Chronic
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic | interventions — molidustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Molidustat (BAY85-3934) (Experimental): Molidustat group
  Interventions: Drug: Molidustat (BAY85-3934)

INTERVENTIONS:
Drug: Molidustat (BAY85-3934) — Starting dose of molidustat once daily (OD) will be titrated based on the subject's Hb (Hemoglobin) response

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Molidustat in dialysis subjects with renal anemia who are not treated with Erythropoiesis-Stimulating Agents (ESAs)

ELIGIBILITY:
Inclusion Criteria:

* Subject with end-stage kidney disease (ESKD) on dialysis (including, hemodiafiltration, hemodialysis, and other modalities except for peritoneal dialysis) weekly or more than weekly
* Body weight > 40 and ≤ 160 kg at screening
* Male or female subject ≥ 20 years of age at screening
* At least one kidney
* Not treated with ESAs and/or HIF-PH inhibitors within 8 weeks prior to randomization. However, in case of the patient washed out from ESAs, when the mean Hb (at least 2 central laboratory measurements must be taken ≥ 2 days apart before dialysis) has decrease to ≥ 0.5 dL from the Hb level (central laboratory measurement, before dialysis) after the last ESA administration, AND the interval from the last ESA administration to the study drug assignment was over 1 week for epoetin-alpha, 2 weeks for darbepoetin alpha or 4 weeks for epoetin beta pegol
* Mean of the last 2 Hb level (central laboratory measurement, before dialysis) during the screening period must be ≥ 8.0 and < 10.0 g/dL (2 measurements must be taken ≥ 2 days apart and the difference between the 2 measurements must be < 1.2 g/dL) with the last screening Hb measurement within 14 days prior to study drug assignment
* Ferritin ≥ 50 ng/mL at screening

Exclusion Criteria:

* New York Heart Association (NYHA) Class III or IV congestive heart failure
* History of cardio- (cerebro-) vascular events (e.g., unstable angina, myocardial infarction, stroke, pulmonary thromboembolism, and acute limb ischemia) within 6 months prior to randomization
* Sustained and poorly controlled arterial hypertension (defined as systolic BP≥ 180mmHg or diastolic BP ≥ 110mmHg) or hypotension (defined as systolic BP < 90mmHg) at randomization
* Proliferative choroidal or retinal disease, such as neovascular age-related macular degeneration or proliferative diabetic retinopathy requiring invasive treatment (e.g., intraocular injections or laser photocoagulation)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2018-10-23 (Actual); Study Completion 2018-11-20 (Actual)

PRIMARY OUTCOMES:
Rate of rise in Hb (Hemoglobin) level (g/dL/week) | Up to 8 weeks
Responder rate: proportion of responders among the subjects | Week 21 to 24
  Responder is defined as meeting all of the following criteria:
  (i) Mean of the Hb levels in the target range (ii) ≥ 50% of the Hb levels in the target range (iii) No rescue treatment

SECONDARY OUTCOMES:
Rate of rise in Hb (Hemoglobin) level (g/dL/week) | Up to 4 weeks
Proportion of subjects who meet each component of the response | Week 21 to 24
  Response:
  (i) Mean of the Hb levels in the target range (ii) ≥ 50% of the Hb levels in the target range (iii) No rescue treatment
Cumulative proportion of subjects who achieve the lower limit of the target Hb range at least once at each visit | Up to 24 weeks
Hb level | Baseline and up to 24 weeks
Change in Hb level | Baseline and up to 24 weeks
Proportion of subjects whose mean hemoglobin levels are above the target range during the evaluation period | Week 21 to 24
Proportion of subjects whose mean hemoglobin levels are below the target range during the evaluation period | Week 21 to 24
Proportion of subjects whose mean hemoglobin levels are in the target range during the evaluation period | Week 21 to 24
Proportion of subjects with hemoglobin levels above the target range | Up to 24 weeks
Proportion of subjects with hemoglobin levels below the target range | Up to 24 weeks
Proportion of subjects with hemoglobin levels in the target range | Up to 24 weeks
Proportion of subjects whose maximum rise in Hb between each consecutive visits is above 0.5 g/dL/week | Up to 24 weeks
  Defined as change in Hb level / duration between two visits (weeks)
Number of participants with serious adverse events | Up to 24 weeks
Maximum concentration (Cmax) of Molidustat | Baseline, Week 8, Week16 and Week 24
Area under the concentration-time curve (AUC) of Molidustat | Baseline, Week 8, Week16 and Week 24
EPO (Erythropoietin) serum concentration of Molidustat | Baseline, Week 8, Week16 and Week 24

CONTACTS AND LOCATIONS:
Locations (20):
- Japan (20):
  - Houshikai Kano hospital, Kasuya-gun, Fukuoka
  - Matsunami General Hospital, Hashima-gun, Gifu
  - Asahikawa-Kosei General Hospital, Asahikawa, Hokkaido
  - Ishikari Hospital, Ishikari, Hokkaido
  - Itami Kidney Clinic, Noboribetsu, Hokkaido
  - Souen Central Hospital, Sapporo, Hokkaido
  - Takasago Seibu Hospital, Takasago, Hyōgo
  - Japanese Red Cross Koga Hospital, Koga, Ibaraki
  - Mito Kyodo General Hospital, Mito, Ibaraki
  - Tokiwa Clinic, Totte, Ibaraki
  - Tsuchiura Beryl Clinic, Tsuchiura, Ibaraki
  - Kikuchi Medical Clinic, Tsukuba, Ibaraki
  - Japanese Red Cross Ishinomaki Hospital, Ishinomaki, Miyagi
  - Iida Hospital, Iida, Nagano
  - Toyonaka Keijinkai Clinic, Toyonaka, Osaka
  - Kodaira Kitaguchi Clinic, Kodaira, Tokyo
  - Medical corporation association Shunshin-kai Inage hospital, Chiba
  - Fukuoka Renal Clinic, Fukuoka
  - Ohmiya Chuo General Hospital, Saitama
  - Yamagata Tokushukai Hospital, Yamagata

REFERENCES:
- [Derived] Akizawa T, Nobori K, Matsuda Y, Hayashi Y, Hayasaki T, Yamamoto H. Molidustat for anemia correction in Japanese patients undergoing hemodialysis: a single-arm, phase 3 study. Ther Apher Dial. 2021 Dec;25(6):917-925. doi: 10.1111/1744-9987.13627. Epub 2021 Mar 22. PMID 33506635
- [Derived] Akizawa T, Taguchi M, Matsuda Y, Iekushi K, Yamada T, Yamamoto H. Molidustat for the treatment of renal anaemia in patients with dialysis-dependent chronic kidney disease: design and rationale of three phase III studies. BMJ Open. 2019 Jun 14;9(6):e026602. doi: 10.1136/bmjopen-2018-026602. PMID 31203241
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/